CLINICAL TRIAL: NCT05849389
Title: Vosoritide for Treatment of Short Stature in Girls With Turner Syndrome
Brief Title: Vosoritide for Short Stature in Turner Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roopa Kanakatti Shankar, MBBS, MS (Other)
Responsible Party: Sponsor-Investigator, Roopa Kanakatti Shankar, MBBS, MS, Director, Turner Syndrome Program, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY0000567
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Turner Syndrome; Short Stature
Keywords: Turner syndrome; Short Stature; Vosoritide
MeSH Terms: conditions — Turner Syndrome; Dwarfism | interventions — vosoritide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vosoritide treatment arm (Experimental): Vosoritide will be administered daily via subcutaneous injection for 12 months using the FDA approved weight-based dosing band strategy for achondroplasia.
  Interventions: Drug: Vosoritide

INTERVENTIONS:
Drug: Vosoritide — Vosoritide administered daily via subcutaneous injection for 12 months using the FDA approved weight-based dosing band strategy for achondroplasia.
  Other Names: Voxzogo

SUMMARY:
Turner syndrome (TS) is characterized by a missing whole or part of the second sex chromosome in a phenotypic female, resulting in short stature due to haploinsufficiency of the short-stature homeobox-containing (SHOX) gene. Growth hormone (GH) is an approved therapy for this condition, although not associated with GH deficiency, and benefits are modest. Vosoritide, a C-type natriuretic peptide (CNP) analog, targets chondrocytes within the growth plate leading to increased cell proliferation and hypertrophy. We hypothesize that patients with TS and short stature will respond to vosoritide treatment leading to increased growth velocity. This study will enroll pre-pubertal girls with TS who are either naïve to GH or have had a poor response to GH therapy. All subjects will be treated with vosoritide for 12 months and will be assessed for safety monitoring and improvement in height outcomes. Annualized growth velocity (AGV) on vosoritide will be compared to AGV in the 6-18 months prior to initiation of vosoritide based on historical data available in the medical record. Subjects with a positive response to therapy will be given the option to continue in the extension phase of the study during which they will continue to receive vosoritide until growth cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s) or guardian(s) are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure. Also, subjects under the age of 18 are willing and able to provide assent (if required) after the nature of the study has been explained and prior to performance of any research-related procedure.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age >3 years 0 days AND <10 years 364 days
4. Pre-pubertal defined as Tanner Stage 1 breasts in females.
5. Patient height <-2 SDS. All height SDS values are calculated using the CDC growth charts/data tables.
6. Patients must have a confirmed diagnosis of Turner Syndrome based on a karyotype with a minimum of 30 cells or on a chromosomal microarray. Subjects with Turner Syndrome mosaicism (such as a 46,XX/45,X karyotype) must have a minimum of 10% mosaicism of 45,X cell line in order to participate in the study.
7. Subjects must either be naïve to growth hormone or have a poor response to growth hormone therapy defined as either:

   1. Subjects completed at least one year of treatment with GH and first year height velocity (HV) below -1 SD according to the National Cooperative Growth Study TS 1st year response to growth hormone height velocity curve.
   2. Subjects receiving GH for more than a year with AGV in the last 6 months < 50%ile for US girls for age/sex). Subjects meeting this criterion are no longer showing catch up growth and may benefit from an alternative form of therapy.

Exclusion Criteria:

1. Growth plate fusion - Defined as a bone age via the Greulich and Pyle method of 13 years. These patients have limited remaining growth potential.
2. Concomitant treatment with growth hormone or recombinant insulin-like growth factor-1 (IGF-1). Patients may have been previously treated with growth hormone or IGF-1 therapy. If the patient is currently on one of these therapies, they will be required to discontinue at least 1 week prior to the screening visit. That decision will be deferred to their treating clinical endocrinologists in conjunction with the patient's guardians. We anticipate that only patients who are having a poor response to their therapy will be interested in enrolling in the current study as there is no rationale for a patient who is receiving growth hormone therapy and having a positive response to enroll in the current study.
3. Prior or concomitant treatment with any form of estrogen, gonadotropin-releasing hormone (GnRH) analog, aromatase inhibitor or oxandrolone
4. History of any type of malignancy
5. Subjects known to have Y-chromosome material unless they have undergone gonadectomy and have fully external female genitalia
6. Chronic medical condition known to affect growth including but not limited to:

   A. Cystic fibrosis B. Diabetes C. Inflammatory Bowel Disease D. Untreated Celiac Disease - If a subject has been diagnosed with celiac disease and has been on a gluten free diet for >12 months and has a tissue transglutaminase antibody within the normal range at screening, then they are eligible for the trial.

   E. Asthma requiring a daily inhaled steroid dose > 400 micrograms of inhaled budesonide per day or equivalent F. Taking daily oral glucocorticoids for any reason G. Note - Attention Deficit hyperactivity Disorder (ADHD) treated with a stimulant and treated hypothyroidism with a normal thyroid stimulating hormone (TSH) will NOT exclude the subject from participating in the trial. Subjects on either stimulant medication or thyroid hormone replacement must be on a stable dose for 3 months prior to the screening visit.

   H. Congenital heart disease which places the subject at increased risk of an adverse cardiac outcome in the setting of hypotension including but not limited to: hypertrophic cardiomyopathy, aortic stenosis with peak gradient >50mmHg, severe aortic regurgitation (defined as pressure half time >500ms by echocardiogram), coronary insufficiency, or any anatomy with a need for an afterload reducing agent. Any patient with baseline abnormalities on echocardiogram will be reviewed with a pediatric cardiologist for appropriateness for inclusion in the study.
7. Malnutrition - Defined as a BMI <5th percentile (CDC growth charts)
8. Any clinically significant abnormality on screening tests as determined by the principal investigator. Abnormal screening labs may be repeated up to 3 months after the screening visit. If those labs are normal on repeat, the subject may proceed into the trial.
9. Known or suspected allergy to trial medication, excipients, or related products
10. The receipt of any investigational drug within 90 days prior to this trial

Ages: 3 Years to 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 12 months
  Number of treatment-emergent adverse events or serious adverse events per study participant
Change from baseline in annualized growth velocity | 12 months
  To evaluate the change from baseline in annualized growth velocity after 12 months of daily subcutaneous injections of vosoritide
Change from baseline in age-sex standardized height standard deviation score | 12 months
  To evaluate the change from baseline in age-sex standardized height standard deviation score (SDS) after 12 months of daily subcutaneous injections of vosoritide

SECONDARY OUTCOMES:
Changes in seated height ratio | 12 months
  To evaluate the seated height ratio as a measure of body proportions compared to baseline after daily subcutaneous injections of vosoritide
Changes in arm span minus standing height | 12 months
  To evaluate the arm span minus standing height as a measure of body proportion compared to baseline after daily subcutaneous injections of vosoritide
Change in Bone Age | 12 months
  To evaluate changes from baseline in bone age/chronological age after 12 months of daily subcutaneous injections of vosoritide

CONTACTS AND LOCATIONS:
Overall Officials: Roopa Kanakatti Shankar, MBBS, MS, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No